CLINICAL TRIAL: NCT07184528
Title: PATCHVALVE Trial: A Prospective Evaluation of Blood Patch and Endobronchial Valves for Persistent Air Leaks - Pilot Study
Brief Title: PATCHVALVE: Endobronchial Valves Plus Blood Patch for Persistent Air Leaks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jason A Beattie, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000315
Record Dates: First submitted 2025-08-25; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Persistent Air Leaks
Keywords: persistent air leaks; Endobronchial Valves; Spiration Valve System; Endobronchial Blood Patch; Intrabronchial Valves
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Bronchoscopic Endobronchial Valve and Blood Patch Treatment Group for Persistent Air Leak Management (Experimental): This study will enroll patients with persistent air leaks (PAL) following lung resection or unrelated to lung resection, who have ipsilateral chest tubes in place and are either not suitable candidates for surgical intervention or have declined surgery. Participants will undergo a combined bronchoscopic approach involving endobronchial valve (EBV) placement and endobronchial blood-patch application, aiming to effectively manage air leaks through a minimally invasive, nonsurgical technique.
  Interventions: Device: Endobronchial Blood Patch; Device: Spiration Valve System (SVS) Placement

INTERVENTIONS:
Device: Endobronchial Blood Patch — This component of the procedure involves sealing persistent air leak (PAL) defects using autologous blood delivered via a balloon catheter. After identifying the target segment, carefully noting the airway angle and distal carina, a sizing balloon is deployed and inflated to ensure a tight seal. Under anesthesia, 30 mL of fresh blood is prepared and infused into the target airway until either visible extravasation occurs or the full volume is delivered. Following this, up to 10 mL of tranexamic acid (TXA) may be administered, again until extravasation occurs or the volume is fully instilled. The balloon remains inflated for 3-5 minutes after the instillation to allow clot formation and sealing of the defect.
Device: Spiration Valve System (SVS) Placement — Once the blood patch component is complete and the balloon is deflated, a Spiration Valve System (SVS) is placed proximally in the airway. The valve acts as a one-way device that decompresses the targeted lung segment while stabilizing the clot created by the blood patch. This supports durable resolution of the air leak, particularly in cases where collateral ventilation might otherwise reduce the efficacy of valve therapy alone.

SUMMARY:
The goal of this study is to evaluate the real-world safety and effectiveness of combining endobronchial valve (IBV) placement with endobronchial blood patching (EBP) for the treatment of persistent air leaks (PALs) in adult patients undergoing bronchoscopy. PALs are a challenging condition often associated with prolonged hospital stays, increased morbidity, and delayed recovery.

The main questions this study aims to answer are:

* Does the combination of endobronchial valve placement and endobronchial blood patching accelerate resolution of persistent air leaks?
* What are the procedural outcomes, complications, and hospital-related metrics (e.g., chest tube duration, length of stay, and readmission rates) associated with this technique?

Participants will:

* Undergo standard-of-care bronchoscopy with identification of air leak source.
* Receive intrabronchial instillation of autologous blood and tranexamic acid (TXA) followed by balloon occlusion and endobronchial valve placement.
* Be followed for resolution of air leak and post-procedure outcomes through standard inpatient monitoring and data collection.

DETAILED DESCRIPTION:
This study will include a prospective cohort of adult patients with persistent air leaks (PALs) undergoing bronchoscopy. The intervention evaluated is a combination approach that includes endobronchial valve placement and instillation of autologous blood with tranexamic acid (TXA), followed by balloon occlusion (referred to as "PATCHVALVE" technique).

Patients will be enrolled and undergo standard imaging and procedural evaluations. For prospective participants, informed consent will be obtained prior to the procedure.

Procedural steps include:

* Identification of the leaking segment using imaging and air leak assessment.
* Instillation of fresh autologous blood (up to 30 mL) followed by TXA (up to 10 mL) via a balloon catheter into the leaking airway segment.
* Balloon occlusion for 3-5 minutes to promote clotting and adherence.
* Deployment of endobronchial valves based on standard criteria.
* Leak reassessment and iterative treatment if necessary.

This study will provide early evidence on the efficacy of this combined approach and help standardize care protocols for managing PALs non-surgically.

ELIGIBILITY:
{Inclusion Criteria}

* Adult (≥18 years) patients who have been diagnosed with persistent air leaks (PALs) due to conditions such as alveolar-pleural fistulas following pulmonary resections, traumatic injury, or underlying lung disease or other cause.
* PAL patients who are deemed non-candidates for surgical intervention or have declined surgery.

{Exclusion Criteria}

* Patients who have received other experimental or investigational treatments for PALs that could confound the results.
* Patients with contraindications to undergoing bronchoscopy, such as severe cardiovascular instability, or those who cannot tolerate the procedure due to other medical reasons.
* Bronchopleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Following Combined Blood Patch and Spiration Valve Application | From enrollment to the end of the observational period at 12 months post-intervention as per standard procedure
  This outcome will assess the safety of the combined blood patch and Spiration valve intervention by measuring the number of participants who experience one or more adverse events. Adverse events may include valve migration, the emergence of new air leaks in lung lobes other than the treated segment, and deterioration in pulmonary function, such as worsened gas exchange or progression to respiratory failure.
  Units: Binary (YES/NO)
Feasibility of Combined Endobronchial Blood Patch and Spiration Valve Procedure | From enrollment to end of procedure.
  Defined as the successful completion of the combined autologous endobronchial blood patch and Spiration Valve procedure.
  Units: Binary (Yes/No - Procedure Completed as Intended)

SECONDARY OUTCOMES:
Change in Air Leak Severity Based on Cerfolio Classification | From enrollment to end of observational period at 12 months post-intervention as per standard procedure
  This refers to the variation or progression in postoperative pulmonary air leaks, categorized based on the Cerfolio classification system. Units: Change in Cerfolio Grade (e.g., Grade 4 to Grade 2)
Time to Air Leak Resolution | From enrollment to end of observational period at 12 months post-intervention as per standard procedure.
  Duration from the onset of a postoperative air leak to its complete cessation. Units: Days
Change in Chest Tube Suction Requirement | From enrollment to end of observational period at 12 months post-intervention as per standard procedure
  This denotes the alteration in the level or need for suction applied to a chest drainage system over time. Units: cmH₂O
Time to Chest Tube Removal | From enrollment to end of observational period at 12 months post-intervention as per standard procedure
  Duration from intervention to successful removal of the chest tube, indicating resolution of the persistent air leak and adequate lung re-expansion. Units: Days
Subsequent Interventions Required Following Blood Patch and Valve Treatment | From enrollment to end of observational period at 12 months post-intervention as per standard procedure
  Incidence and nature of additional therapeutic procedures required to manage persistent air leaks following the initial combined blood patch and valve intervention. Units: Number of participants requiring ≥1 additional intervention
Incidence of Respiratory Infections Following Combined Blood Patch and Spiration Valve Application | From enrollment to the end of the observational period at 12 months post-intervention.
  This outcome will specifically evaluate the number of participants who develop respiratory infections following the intervention. Respiratory infections of interest include post-obstructive pneumonia and other clinically documented respiratory infections potentially related to the procedure.
  Units: Binary (YES/NO)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Beattie, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Isreal Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durrance RJ, D'Souza KG, Obata R, Bradley EC, Perwaiz MK. Endobronchial blood-patch: A novel technique for a persistent pleural air leak. Respir Med Case Rep. 2022 May 28;38:101670. doi: 10.1016/j.rmcr.2022.101670. eCollection 2022. PMID 35656093
- [Background] Watanabe S, Watanabe T, Urayama H. Endobronchial occlusion method of bronchopleural fistula with metallic coils and glue. Thorac Cardiovasc Surg. 2003 Apr;51(2):106-8. doi: 10.1055/s-2003-38981. PMID 12730823
- [Background] Takaoka K, Inoue S, Ohira S. Central bronchopleural fistulas closed by bronchoscopic injection of absolute ethanol. Chest. 2002 Jul;122(1):374-8. doi: 10.1378/chest.122.1.374. PMID 12114386
- [Background] Lopez C, Facciolo F, Lequaglie C, Rendina EA, Saita S, Dell'Amore D, Sollitto F, Urciuoli G, Loizzi M, Cisternino ML, Granone P, Angelelli A, Cardillo G, Mucilli F, Di Rienzo G. Efficacy and safety of fibrin sealant patch in the treatment of air leakage in thoracic surgery. Minerva Chir. 2013 Dec;68(6):559-67. PMID 24193288
- [Background] Thistlethwaite PA, Luketich JD, Ferson PF, Keenan RJ, Jamieson SW. Ablation of persistent air leaks after thoracic procedures with fibrin sealant. Ann Thorac Surg. 1999 Feb;67(2):575-7. doi: 10.1016/s0003-4975(98)01292-2. PMID 10197706
- [Background] Majid A, Kheir F, Sierra-Ruiz M, Ghattas C, Parikh M, Channick C, Keyes C, Chee A, Fernandez-Bussy S, Gangadharan S, Folch E. Assessment of Fissure Integrity in Patients With Intrabronchial Valves for Treatment of Prolonged Air Leak. Ann Thorac Surg. 2019 Feb;107(2):407-411. doi: 10.1016/j.athoracsur.2018.08.046. Epub 2018 Oct 10. PMID 30315804
- [Background] Ding M, Gao YD, Zeng XT, Guo Y, Yang J. Endobronchial one-way valves for treatment of persistent air leaks: a systematic review. Respir Res. 2017 Nov 6;18(1):186. doi: 10.1186/s12931-017-0666-y. PMID 29110704
- [Background] Gillespie CT, Sterman DH, Cerfolio RJ, Nader D, Mulligan MS, Mularski RA, Musani AI, Kucharczuk JC, Gonzalez HX, Springmeyer SC. Endobronchial valve treatment for prolonged air leaks of the lung: a case series. Ann Thorac Surg. 2011 Jan;91(1):270-3. doi: 10.1016/j.athoracsur.2010.07.093. PMID 21172529
- [Background] Mahajan AK, Khandhar SJ. Bronchoscopic valves for prolonged air leak: current status and technique. J Thorac Dis. 2017 Mar;9(Suppl 2):S110-S115. doi: 10.21037/jtd.2016.12.63. PMID 28446973
- [Background] Dugan KC, Laxmanan B, Murgu S, Hogarth DK. Management of Persistent Air Leaks. Chest. 2017 Aug;152(2):417-423. doi: 10.1016/j.chest.2017.02.020. Epub 2017 Mar 4. PMID 28267436
- [Background] Johnson BH, Johnston SS, Tewari P, Afolabi M, Danker Iii W. Clinical and Economic Burden Associated with Prolonged Air Leaks Among Patients Undergoing Thoracic Resection: A Retrospective Database Analysis. Clinicoecon Outcomes Res. 2023 Apr 11;15:269-280. doi: 10.2147/CEOR.S405270. eCollection 2023. PMID 37070065
- [Background] Chee CB, Abisheganaden J, Yeo JK, Lee P, Huan PY, Poh SC, Wang YT. Persistent air-leak in spontaneous pneumothorax--clinical course and outcome. Respir Med. 1998 May;92(5):757-61. doi: 10.1016/s0954-6111(98)90008-7. PMID 9713636
- [Background] Huang X, Ding L, Xu H. Bronchoscopic valve placement for the treatment of persistent air leaks. Medicine (Baltimore). 2018 Mar;97(13):e0183. doi: 10.1097/MD.0000000000010183. PMID 29595651
- [Background] Lazarus DR, Casal RF. Persistent air leaks: a review with an emphasis on bronchoscopic management. J Thorac Dis. 2017 Nov;9(11):4660-4670. doi: 10.21037/jtd.2017.10.122. PMID 29268535